CLINICAL TRIAL: NCT06474702
Title: Predicting Violent Outburst in Inpatient Pediatric Psychiatry Ward Using a Wearable Device.
Status: Not yet recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Doron Gothelf MD, head of child and adolescent psychiatry division, Sheba Medical Center
Other Study IDs: 1135-24-SMC
Record Dates: First submitted 2024-06-17; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Child Behavior Disorders
MeSH Terms: conditions — Child Behavior Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study arm: the investigator will utilize "Fitbit-Charge 4" a wearable 'smart-watch' in order to collect patients' physiological measurements, including continuous heart rate, heart-rate variability and breathing rate, as well as behavioral measurements such as movements and sleep pattern in order to predict aggression and violence outburst in children under 12 years old admitted at an inpatient psychiatric ward and characterization of those physiological measures in the prediction of aggression and violence outbursts.
  Interventions: Device: 'Fitbit charge 4' 'smart-watch'-

INTERVENTIONS:
Device: 'Fitbit charge 4' 'smart-watch'- — smartwatch device that collects physiological measures

SUMMARY:
The investigator will investigate the use of non-invasive wearable device physiological measures. this in order to predict aggression, and violence outburst in children under 12 years old, which are admitted at an inpatient psychiatric ward. also, the investigator will try to do a characterization of those physiological measures in the prediction of aggression and violence outbursts.

ELIGIBILITY:
Inclusion Criteria:

* the investigator will include patients under the age of 13 with various mental disorders admitted to our inpatient psychiatry ward at 'Edmond and Lily Safra' Children's Hospital, Sheba Medical Centre, Tel Hashomer, Ramat Gan, Israel during 2024.

Exclusion Criteria:

* the investigator will exclude patients that were hospitalized but did not want to participate, or couldn't participate due to increased sensorial sensitive to the device. the investigator will exclude patients with no violence outburst or aggressive attitude that were hospitalized at our inpatient psychiatric ward during 2024. additional, patients who suffers dermatological illnesses and might show allergic reactions to the device material on their wrist will be excluded.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with mental ilnesses hospitalized at out inpatient psychiatric ward
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
physiological parameter | 12 months (july 2024-july 2025)
  Heart rate
physiological parameter | 12 months (july 2024-july 2025)
  heart rate variability, the data of heart rate variability is based on respiratory rate (outcome 3) and heart rate (outcome 1)
physiological parameter | 12 months (july 2024-july 2025)
  respiratory rate
physiological parameter | 12 months (july 2024-july 2025)
  sleep patterns, the data of sleep pattern is based on movements (outcome 5) and heart rate (outcome 1)
movements. | 12 months (july 2024-july 2025)
  movements frequency of the patient, collected by the smart-watch using 3 axis-accelerometer that can detect movements in 3 dimensions. for example, number of steps taken.

SECONDARY OUTCOMES:
violence assessment with 'MOAS' score system. | 12 months (july 2024-july 2025)
  using 'MOAS', the Modified Overt Aggression Scale score system filled by the department staff manually on each day and outburst description. the score system is made up of four categories (verbal aggression, aggression against objects, aggression against self, and aggression against others. each category is ranked by numbers. range of total score is between 0-40. higher score usually higher than 20 indicating more aggressive behavior which means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Gothelf, M.D, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No